## Family Check-Up Online for Middle School Parents

November 21st, 2023

## Family Check-Up Online for Middle School Parents Parent/Guardian Consent Form

All parents of youth in grades 6-8 who are enrolled in select public schools are being invited to participate in a free program called "Family Check-Up Online for Middle School Parents". This project is being conducted by Dr. Dustin Pardini at Arizona State University using funding provided by the Arizona Health Care Cost Containment System and Arizona State University. The goal of this program is to help parents identify existing family strengths and learn about different parenting strategies that have been shown to improve family functioning and promote positive adolescent health and emotional/behavioral wellness. The program involves completing a series of five interactive modules online which you can access using any internet connected device. Each online module takes ~15-20 minutes to complete and can be done over the course of eight weeks whenever you have free time. During this 8-week period, you are encouraged to revisit the online modules to identify and practice implementing different parenting strategies consistent with your family goals. You will also be assigned to a program staff member whom you may meet with via phone or Zoom at any point for additional support while working through the program. At the end of the 8-week period, you will be able to access an online feedback report module which is designed to show you improvements you have made using the parenting strategies described within each program module.

One of the goals of this project is to determine whether different types of staff support can help improve outcomes for parents completing the Family Check-Up Online program. To address this goal, parents will be randomly assigned to one of two conditions. Parents randomized to the "Informational Support Specialist" condition will be assigned to a staff member who they can meet with via the phone or online using Zoom if they have any questions regarding the content of the program. Parents randomly assigned to the "Guidance Coach" condition will be assigned to a staff member who will invite them to participate in 1-3 brief check-in meetings while completing the program via phone or online using Zoom. These coaching meetings are designed to support parents in completing the program and provide guidance on how to use aspects of the program to meet the goals they have for their family. These meetings can be conducted at a time that works best for you. In order to assess the utility of these different types of support, we will document the number and duration of any meetings you have with program staff, as well as what aspects of the program were discussed. The program website will also collect digital information about your engagement with the Family Check-up Online material, including the number of modules completed and duration of time spent on each module. We will use this information to better understand how parents interact with the program and determine whether parents benefit from receiving different types of staff support.

If you agree to participate, you will first be asked to complete a brief survey (~15-25 minutes) about your current family structure and functioning, including your current parenting practices, feelings, and beliefs; as well as your child's emotions (e.g., stress), behaviors (e.g., arguing), and school performance. Once the survey is completed, you will be emailed a link allowing you to access the Family Check-up Online program, along with contact information for your assigned Informational Support Specialist or Guidance Coach. If you complete all five modules of the program and the online feedback report module at the end of 8-week period, you will be emailed a \$20 Amazon gift card. Three months after you start the program, you will also be emailed a link to access a brief follow-up survey (~15-25 minutes). Questions will be repeated from the first survey to measure changes in family functioning to help improve the program. If you complete this survey, you will be emailed a \$10 Amazon gift card. Additionally, one out of every 25 parents who complete this follow-up survey will also be entered into a drawing to receive a \$50 Amazon gift card.

Participation in this study is voluntary. If you choose not to participate there will be no penalty. You also may stop participating at any time without penalty. This project is also designed to protect your privacy. No one besides select project staff at Arizona State University will have access to any personally identifiable information you provide as part of this project. The information collected as part of this project will be used in summary reports, publications and presentations, and this de-identified information may be shared with other investigators for future research. However, your personally identifiable data (e.g., name, contact information) will never be reported or shared with anyone outside of project staff, and all personally identifiable data collected as part of this project will be permanently destroyed once the project has been completed. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. Individual results and study findings will not be reported back to participants.

There are minimal risks associated with this study. One potential risk is that you may feel uncomfortable with some of the survey questions or material covered as part of the Family Check-up program. However, you may skip any survey questions that you do not want to answer and can withdraw from the program at any time without penalty. Another possible risk is breach of confidentiality. We are committed to protecting your personal information, which will be stored separately from your survey responses and program engagement information. Instead, we will assign you a participant ID

number. All data will be stored on a secure, password-protected computer server. Only limited research staff will have access to this server. However, should you disclose to study staff that a child in your home has experienced abuse or neglect, we are mandated by Arizona law to report these concerns to the Department of Child Safety (see ARS §13-3620).

Parents may experience some benefits from this study. All parents will receive a resource list for support services including local agencies that provide a variety of services (e.g., family behavioral and mental health services, financial support agencies) after completing the initial survey. Although this program is not an FDA approved cure or treatment for any physical/ mental health conditions, families may also find the program to be useful. Research has shown that the program enhances parents' self-confidence that they can implement skills and strategies that promote positive emotional and behavioral health among teens. Parental adoption of the strategies outline in the program may also help protect youth from engaging in risky behaviors during later adolescence (e.g., substance use, delinquency).

This project has been approved by the research review board at ASU. If you have any questions about the project or would like more information about the Family Check-Up program, please contact Dr. Dustin Pardini at <a href="mailto:dpardini@asu.edu">dpardini@asu.edu</a> or 602-496-2357. If you have any questions about your rights as a subject/participant in this research, or if you feel you have been placed at risk, you can contact the Chair of the Human Subjects Institutional Review Board, through the ASU Office of Research Integrity and Assurance, at (480) 965-6788. State that you are calling about the Family Check-Up Online for Middle School Parents study. Someone will return your call as soon as possible.

Please indicate whether or not you consent to participate in the Family Check-Up study.

| YES, I consent to take part in this study. |
|---|
| NO, I do not consent to take part in this study. |
| If yes, please provide the following information. As stated above, this information is only accessible to program staff and will be permanently destroyed once the project has been completed. |
| Your first and last name: |
| Your email address: |
| Your cell phone number: |
| Your street address: |
| Your ZIP code: |
| Your child's district/school that referred you to the program: |
| First name of the child enrolled in grade 6-8 at the school above. If you have more than one child in grade 6-8 attending the school, enter the youngest child's name: |
| What language would you like to use when completing the Family Check-up program? |
| <b>English</b> |
| Spanish Spanish |
| For issues related to the program, is it okay for project staff to leave a voicemail? |
| Yes |
| No No |
| For issues related to the program, is it okay for project staff to contact you via text? Yes |
| No No |
| Do you use WhatsApp for calling/texting? Yes |
| □ No |

| What days and times would typically work best for you to meet with a program coach? Weekday Mornings |
|---|
| Weekday Afternoons |
| Weekday Evenings |
| Weekends |